CLINICAL TRIAL: NCT03096977
Title: Use of the Nine Holes Peg Test in Multiple Sclerosis: Participation of Elementary Neurological Components in the Functional Evaluation of Manual Dexterity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Bernard Dachy, Head of Clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUB-Nine Holes Peg Hands
Record Dates: First submitted 2017-03-24; First posted 2017-03-31 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: Hand dexterity; Multiple sclerosis; Nine Holes Peg
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHUB-TST02 patients (Experimental): All patients who participated in the NCT02805634 (CHUB-TST02) study.
  Interventions: Diagnostic Test: Scale for the assessment and rating of ataxia (SARA); Device: JAMAR hand dynamometer; Device: Vibratory sensibility testing; Device: Sermes and Weinstein test; Device: Weber test

INTERVENTIONS:
Diagnostic Test: Scale for the assessment and rating of ataxia (SARA) — Clinical evaluation of the manual dexterity through the SARA scale.
Device: JAMAR hand dynamometer — Clinical evaluation of the prehension force using a JAMAR Dynamometer.
  The prehension effort is made with the arm along the body, forearm horizontal, elbow flexed at 90 degrees, wrist in neutral position. The handle of the dynamometer is set to the second notch. The effort required is maximum effort.
  Verbal encouragement is given during four successive tentative: the last three are averaged.
  Each effort will be separated by a rest period of one minute. Interval: 1 min - Repeat: 3 times per hand
Device: Vibratory sensibility testing — Test carried out using a tuned fork applied to the styloid radial process.
  Position of the evaluated: elbow to the body with forearms horizontal and the wrist in neutral position. Stimulate the tuning fork and apply it to the styloid process of the radius. Ask the patient to say when he no longer feels the vibration.
  Repeat 3 times for each hand.
Device: Sermes and Weinstein test — Instrumental, quantitative method of tactile pressure sensation (dermal contact at constant pressure) using monofilaments. The monofilaments bend when a threshold force is applied to them.There is a kit of 5 monofilaments, each one corresponding to a different functional level.
  Familiarize the patient with the test, eyes open, on a normal healthy side. Determine the level of perception of the healthy side, eyes closed. Start with the finest monofilament. If the answer is negative, go to the next monofilament.
  The monofilaments applications are randomly made in the Wynn Parry areas, 3 times / area for blue and green filaments, then 1 time / zone for others.
  The monofilament must be applied in 1.5 sec, held 1.5 sec, removed in 1.5 sec. The patient must give a verbal response "yes" when he perceives the contact and the response time must be less than 3 sec.
Device: Weber test — Evaluate the discrimination of 2 motionless points. The tactile discrimination threshold is the smallest distance separating 2 simultaneous stimulations that are located and perceived separately.
  The pressure stops at the whitening of the skin. The patient should specify if he feels one or two spikes.
  To determine the discrimination threshold:
  Perform 10 stimulations of the same spacing in the same area. The smallest interval for which 7 correct answers are obtained is retained as threshold value.
  Perform the test 3 times.

SUMMARY:
This study lies in the continuity of the study with identification number NCT02805634. It will be performed on the same group of patients and will aim to assess the manual dexterity, in order to better assign kinesitherapy treatments and increase the utilisation capacity of the hand.

ELIGIBILITY:
Inclusion Criteria:

* All patients included in the NCT02805634 study

Exclusion Criteria:

* None

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Scale for the assessment and rating of ataxia (SARA) | 1 year
  Scale for the assessment and rating of ataxia (SARA)
Prehension force | 1 year
  Prehension force, using a JAMAR hand dynamometer
Tuned fork result | 1 year
  Vibratory sensibility testing
Sermes and Weinstein test | 1 year
  Tactile pressure sensation testing
Weber test | 1 year
  Evaluate the discrimination of 2 motionless points

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Dachy, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No